CLINICAL TRIAL: NCT00843063
Title: Famotidine vs. Pantoprazole to Prevent Recurrent Aspirin-Induced Peptic Ulcer/Erosion - a Randomized Controlled Study
Brief Title: Famotidine Compared With Pantoprazole to Prevent Recurrent Aspirin-Induced Peptic Ulcer/Erosion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ruttonjee Hospital (Other)
Responsible Party: Dr Fook Hong Ng, Ruttonjee Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HKEC 2004-016
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Peptic Ulcer/Erosions
Keywords: pantoprazole; famotidine; aspirin; dyspepsia; gastrointestinal bleeding; peptic ulcer / erosion
MeSH Terms: conditions — Peptic Ulcer; Dyspepsia; Gastrointestinal Hemorrhage | interventions — Famotidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pantoprazole (Active Comparator): pantoprazole 20 mg om and matching placebo nocte
  Interventions: Drug: pantoprazole vs famotidine
- famotidine (Active Comparator): Famotidine 40 mg om and nocte
  Interventions: Drug: pantoprazole vs famotidine

INTERVENTIONS:
Drug: pantoprazole vs famotidine — pantoprazole 20 mg om and matching placebo nocte vs. famotidine 40 mg om and nocte
  Other Names: pantoloc; famotidine

SUMMARY:
Low-dose aspirin can prevent cerebral and cardiovascular accidents in individuals with symptomatic atherothrombotic disease, but its use is frequently limited by gastrointestinal side effects.

The position of H2-receptor antagonists as a step-down therapy after healing of peptic ulcer or erosions by proton pump inhibitor is unclear.

The objective of this randomized, double blinded control study was to compare the efficacy of high-dose famotidine with pantoprazole in the prevention of recurrent dyspeptic or complicated ulcer/ erosions in patients taking low-dose aspirin

DETAILED DESCRIPTION:
Low-dose aspirin can prevent cerebral and cardiovascular accidents in individuals with symptomatic atherothrombotic disease . Its use is frequently limited by gastrointestinal side effects, ranging from dyspepsia (31%) to life-threatening bleeding or perforation of gastroduodenal ulcers (3.1%) over a period of 4 years .

The best approach for the secondary prevention of low-dose aspirin induced symptomatic peptic ulcer or erosions in patients who need to continue aspirin remain uncertain. At present, eradication of Helicobacter pylori infection and long-term maintenance with proton pump inhibitor PPI appears to be the best options.

The position of H2-receptor antagonists (H2RA) as a step-down therapy after healing of peptic ulcer or erosions is unclear.

The objective of this randomized, double blinded control study was to compare the efficacy of high-dose famotidine with pantoprazole in the prevention of recurrent dyspeptic or complicated ulcer/ erosions in patients taking low-dose aspirin.

ELIGIBILITY:
Inclusion Criteria:

* upper GIB or dyspepsia due to peptic ulcers / erosions while receiving low-dose aspirin with a daily dose ranging from 80 mg to 320 mg
* endoscopy revealed a gastric or duodenal ulcers of 3 mm or more in diameter with unequivocal depth, or more than 5 erosions in the stomach or duodenum
* they required continuous low-dose aspirin for the secondary prevention of coronary heart disease, peripheral vascular disease and ischemic stroke or transient ischemic attacks
* 18 years old or older.

Exclusion Criteria:

* concurrent erosive or ulcerative esophagitis
* pyloric stenosis
* previous gastric or duodenal surgery other than oversewing of a perforation
* thrombocytopenia
* renal failure with estimated creatinine clearance less than 10 ml / min
* active cancer
* known allergic to aspirin, famotidine or pantoprazole
* pregnancy, lactation, child-bearing potential in the absence of contraception
* psychosomatic disorder
* planned co-prescription of nonsteriodal anti-inflammatory drugs corticosteriod, or anticoagulant
* disorders that might modify the absorption of study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2004-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The primary end-point was the recurrence of dyspeptic or complicated ulcer / erosions. | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fook Hong Ng, M.D., Principal Investigator — Department of Medicine, Ruttonjee Hospital
Locations (1):
- Ruttonjee Hospital, Wan Chai, Hong Kong, China